CLINICAL TRIAL: NCT01889979
Title: Tramadol for Labour Analgesia in Low Risk Primiparous Women. Double Blind, Randomized, Controlled Trial.
Brief Title: Tramadol for Labour Analgesia in Low Risk Primiparous Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Saint Thomas Hospital, Panama (Other)
Responsible Party: Principal Investigator, Osvaldo A. Reyes T., Coordinator of Research, Saint Thomas Hospital, Panama
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MHST2012-09
Record Dates: First submitted 2013-06-26; First posted 2013-07-01 (Estimated); Last update posted 2013-07-09 (Estimated); Status verified 2013-07

CONDITIONS: Pain During Labour
Keywords: Pain during labour; Duration of labour; Apgar score; Umbilical cord pH
MeSH Terms: interventions — Tramadol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tramadol (Experimental): 100 mg of tramadol SC (single dose) = 2 mL
  Interventions: Drug: Tramadol
- Placebo (Placebo Comparator): 2 mL of a sterile solution SC
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tramadol — 100 mg of Tramadol was applied in the forearm SC (single dose).
  Arms: Tramadol
Drug: Placebo — 2 ml of a sterile solution was applied in the forearm SC (single dose).
  Arms: Placebo

SUMMARY:
Tramadol is a centrally acting synthetic analgesic used to treat moderate to moderately severe pain. It has been previously evaluated as a method to reduce pain during labour, but there is always some fear related to its effects (neonatal respiratory depression). The purpose of our study was to evaluate the efficacy of subcutaneous tramadol in regards to pain during labour, duration of labour and neonatal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age between 37 and 40 6/7 weeks
* Primiparous patient
* Singleton
* 4 to 5 cms of dilation
* Intact membranes or spontaneous rupture of membranes less than 2 hours
* Fetus in a vertex presentation
* Gynecoid pelvis by clinical examination

Exclusion Criteria:

* Multiparous
* Multiple pregnancies
* Any pathology
* Induction of labour with prostaglandins

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-10; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Pain during labour | 6 hours
  Pain during labour was evaluated using the Visual Analogue Scale during the first six hours after the application of the drug (tramadol or placebo).

SECONDARY OUTCOMES:
Duration of labour | 12 hours
  The duration of labour in minutes (all patients were admitted with 4-5 cms of dilation), comparing both groups.
Neonatal outcomes | 48 hours
  Apgar score at minute one and five and umbilical cord pH were evaluated and compared between both groups.
Side effects | 48 hours
  Maternal respiratory depression, headaches, nausea and dizziness were evaluated in both groups.
Requirements of oxytocin | 12 hours
  Maximum dose of oxytocin (mU/min) required to have regular uterine contractions.

CONTACTS AND LOCATIONS:
Overall Officials: Osvaldo Reyes, MD, Principal Investigator — Saint Thomas Maternity Hospital; Riggie Castillo, MD, Principal Investigator — Saint Thomas Maternity Hospital
Locations (1):
- Saint Thomas Maternity Hospital, Panama City, Panama